CLINICAL TRIAL: NCT06017869
Title: PHASE II, OPEN LABEL, SINGLE DOSE STUDY OF THE SAFETY AND EFFICACY OF MNV-201 FOR THE TREATMENT OF PEARSON SYNDROME
Brief Title: Evaluate the Safety and Therapeutic Effects of a Single Intravenous Infusion (IV) of Autologous CD34+ Cells Enriched With Allogenic Placenta-derived Mitochondria in Patients With a Diagnosis of Pearson Syndrome (PS)
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Minovia Therapeutics Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MNV-010
Record Dates: First submitted 2023-08-24; First posted 2023-08-30 (Actual); Last update posted 2025-06-22 (Actual); Status verified 2025-05

CONDITIONS: Mitochondrial Diseases; Pearson Syndrome
Keywords: Autologous; Mitochondrial; Pearson; Transplantation; Stem cell
MeSH Terms: conditions — Mitochondrial Diseases; VLCAD deficiency

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Autologous CD34+ cells enriched with allogenic placenta-derived mitochondria (Experimental)
  Interventions: Biological: MNV-201

INTERVENTIONS:
Biological: MNV-201 — Autologous CD34+ cells are isolated from the participant's peripheral blood after mobilization by leukapheresis. Allogeneic mitochondria are isolated under aseptic conditions from healthy donor placenta, cryopreserved and qualified before use.
  Other Names: CD34+ cells enriched with allogeneic placenta derived mitochondria

SUMMARY:
Primary Mitochondrial diseases are a clinically and genetically heterogeneous group of disorders caused by mutations in genes encoded by nuclear Deoxyribonucleic Acid (DNA) or by mutations and/or deletions in the mitochondrial DNA (mtDNA). While some mitochondrial disorders only affect a single organ (e.g., the eye in Leber hereditary optic neuropathy [LHON]), many involve multiple organs. Mitochondrial disorders may present at any age and a frequent feature is the increasing number of organs involved in the course of the disease.

Minovia Therapeutics Ltd. ("Minovia") is a biotech company developing novel therapeutics based on its mitochondrial augmentation technology (MAT). MNV-201 is a cell therapy produced by MAT that consists of the participant's autologous CD34+ hematopoietic stem and progenitor cells (HSPCs) enriched with allogeneic placental-derived mitochondria, manufactured in Minovia's GMP facility.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female participants aged from 1 to 18 years old.
2. Diagnosis of Pearson Syndrome (current or history) as verified by molecular identification of deletion in mtDNA of peripheral blood. Participants are diagnosed with PS Participant can be in either the PS manifestations of the disease or may have transitioned to Kearns Sayre Syndrome (KSS) manifestations but has a history of PS.
3. Participants have failure to thrive (height SDS smaller than -1)
4. Participants should have at least 12 months' history of body weight and height and calculated GFR (from creatinine) before treatment.
5. Body weight ≥ 10 kg.
6. Participants' living parent(s) and/or legal guardian(s) able to understand and provide voluntary written informed consent.
7. Participants' parents or legal guardian have a good understanding of the study and nature of the procedure and are expected to be able to comply with study visit schedules and caregiver assessments without difficulty.
8. Participants' parents or legal guardian provides written informed consent prior to study participation.
9. Participants are medically able to undergo the study interventions as determined by the Investigator.

Exclusion criteria:

1. History of infection with HIV-1, HIV-2, or HTLV I/II.
2. Participants have any active infection.
3. Participants have been diagnosed with Myelodysplastic Syndrome, by FISH and/or karyotype.
4. Participants are unable to undergo apheresis.
5. Participants have known hypersensitivity to murine proteins or iron-dextran.
6. Participants have severe chronic infection.
7. Participants have disease or conditions that may risk the participant or interfere with the ability to interpret the study results.
8. History of malignancy.
9. History of treatment with gene therapy, allogeneic bone marrow or cord blood transplantation.
10. Participants have had a change in growth hormone regimen in less than 2 years prior to treatment.
11. Participants have participated in another clinical trial or received other experimental medications outside a clinical trial within 1 month prior to start of this study.
12. Participants who are pregnant or intend to become pregnant in the next 12 months.
13. In the opinion of the Investigator, the participant is unsuitable for participating in the study for any reason.

Ages: 1 Year to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 6 (Estimated)
Dates: Start 2023-07-31 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
Occurrence of treatment-related adverse events | 12 months post treatment.
  Occurrence of treatment-related adverse events as assessed by CTCAE v5.0 following MNV-201 infusion
Height SDS | 24 months
  Improvement from baseline to 12 months post treatment in height SDS compared to the calculated change in height SDS in the 12 months prior to treatment.

SECONDARY OUTCOMES:
Height SDS | 12 months
  Improvement from baseline to 6 months post treatment in height SDS compared to the calculated change in height SDS in the 6 months prior to treatment.
Calculated GFR Slope | 24 months
  Improvement in calculated GFR slope 6- and/or 12-months post treatment relative to 6 and/or 12 months prior to treatment (respectively)

OTHER OUTCOMES:
Exploratory endpoint: Organ dysfunction | 24 months
  Improvement in any of the measurements below of organ dysfunction at 6- and/or 12-month post-treatment compared to Baseline
  * Renal glomerulopathy measured by level of cystatin-C or creatinine
  * Renal tubulopathy measured by urine amino acids
  * Renal tubulopathy measured by blood bicarbonate
  * Gastrointestinal activity measured by albumin
  * Gastrointestinal activity measured by pediatric PedsQL 3.0 Gastrointestinal Symptoms Module
  * Pancreas activity measured by insulin
  * Pancreas activity measured by C-peptide
  * Heart activity measured by ECG
  * Growth measured by GDF15
  * Growth measured by IGF1
  * Growth measured by IGFBP
  * Change in physician organ involvement score (see appendix C)
  * Renal glomerulopathy measured by slope of change in eGFR calculated from cystatin-C at 6- or 12-month post-treatment compared to that calculated in the 6- or 12- month period prior to baseline.
Exploratory endpoint: IPMDS | 12 months
  Improvement from baseline in normalized International Pediatric Mitochondrial Disease Scale (IPMDS) scores (total score or each of three separate components) at 6- or 12-month post-treatment compared to Baseline.
Exploratory endpoint: Frequency of Hospitalizations | 24 months
  Reduction in frequency of hospitalization(s) during the 6- and/or 12-months post treatment relative to the 6 and/or 12 months (respectively) prior to treatment
Exploratory endpoint: Length of Hospitalizations | 24 months
  Reduction of length of hospitalization(s) during the 6- and/or 12-months post treatment relative to the 6 and/or 12 months (respectively) prior to treatment.
Exploratory endpoint: exogenous mtDNA | 12 months
  Pharmacokinetic measurements: exogenous mtDNA analysis in PBMCs at 6- and/or 12-month time points
Exploratory endpoint: Blood based biomarkers | 12 months
  Change in blood-based biomarkers at 6- and/or 12-month post-treatment compared to Baseline
  * Mitochondrial quantity and activity (full length mtDNA copy number in PBMC and/or whole blood); ATP content of PBMCs;
  * Anti-mitochondrial antibody level
  * PBMC subset analysis.
Exploratory endpoint: Height SDS | 12 months
  Improvement in height SDS at 6 and/or 12 months relative to natural history available (prospective and/or retrospective)
Exploratory endpoint: weight SDS | 24 months
  Improvement in weight SDS in 6-month and/or 12-month period after treatment relative to 6- and/or 12-month period (respectively) prior to treatment.

CONTACTS AND LOCATIONS:
Locations (1):
- Sheba Medical Center, Ramat Gan, Israel, Israel

IPD SHARING:
Plan to Share IPD: No